CLINICAL TRIAL: NCT05720988
Title: Tagraxofusp-Based Therapy to Eradicate Measurable Residual Disease of Acute Myelogenous Leukemia Prior to Allogeneic Hematopoietic Cell Transplantation
Brief Title: Tagraxofusp to Eradicate Measurable Residual Disease in Patients With Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: trial was not opened
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-001115; NCI-2021-12912 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-01-11; First posted 2023-02-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (tagraxofusp-erzs) (Active Comparator): Patients receive tagraxofusp-erzs IV QD over 15 minutes on days 1-5. Treatment repeats every 28-42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Tagraxofusp-erzs
- Cohort II (azacitidine, tagraxofusp-erzs) (Experimental): Patients receive azacitidine SC daily on days 1-5 and tagraxofusp-erzs IV QD over 15 minutes on days 8-12. Treatment repeats every 28-42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Biological: Tagraxofusp-erzs

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: Cohort II (azacitidine, tagraxofusp-erzs)
Biological: Tagraxofusp-erzs — Given IV
  Other Names: Diphtheria Toxin(388)-Interleukin-3 Fusion Protein; DT(388)-IL3 Fusion Protein; DT388IL3 fusion protein; Elzonris; IL3R-targeting Fusion Protein SL-401; SL-401; Tagraxofusp; Tagraxofusp ERZS

SUMMARY:
This phase Ib/II trial tests the safety of tagraxofusp when given with or without azacitidine in patients with acute myeloid leukemia in remission with measurable residual disease who will undergo allogeneic hematopoietic cell transplant. Tagraxofusp is a recombinant protein consisting of IL-3 conjugated to a truncated diptheria toxin. The IL-3 attaches to the cancer cells and the toxic substance kills them. Azacitidine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Tagraxofusp and azacitidine may work better to kill cancer cells and eradicate measurable residual disease in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of tagraxofusp-erzs (tagraxofusp) with or without azacitidine in participants with acute myeloid leukemia (AML) in remission who are planned to undergo allogeneic hematopoietic cell transplantation (alloHCT).

SECONDARY OBJECTIVES:

I. To estimate the rate of conversion from measurable residual disease (MRD) positive (>= 0.01% by multiparametric flow cytometry [MPFC]) pre-investigational therapy to MRD negative (=< 0.01% by MPFC) after 1 or 2 cycles of investigational therapy.

II. To estimate the rate of conversion from MRD positive (>= 0.01% by MPFC) pre-investigational therapy to MRD negative (=< 0.01% by MPFC) post-investigational therapy within 30 days prior to initiation of transplant conditioning regimen and at day +100 following alloHCT.

III. To evaluate if adverse effects of this investigational combination leads to delays in alloHCT.

IV. To evaluate if this investigational therapy results in liver toxicities after alloHCT such as sinusoidal obstruction syndrome.

V. To evaluate relapse rate following alloHCT in participants who receive investigational therapy.

VI. To evaluate MRD progression following alloHCT in participants who receive investigational therapy.

VII. To evaluate 1-year survival following alloHCT in participants who receive investigational therapy.

EXPLORATORY OBJECTIVES:

I. To estimate the rate of conversion from MRD positive to MRD negative by means of next generation sequencing.

II. To describe the level of CD123 expression on leukemia blasts in the bone marrow specimen at diagnosis and/or time of relapse and the association with achievement of MRD negativity post-investigational therapy.

III. To evaluate the number of days to full donor T-cell chimerism following alloHCT.

OUTLINE: This is a dose-escalation study of tagraxofusp-erzs . Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive tagraxofusp-erzs intravenously (IV) once daily (QD) over 15 minutes on days 1-5. Treatment repeats every 28-42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive azacitidine subcutaneously (SC) daily on days 1-5 and tagraxofusp-erzs IV QD over 15 minutes on days 8-12. Treatment repeats every 28-42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* AML in first or second remission, including:

  * Complete remission (CR), defined as bone marrow blasts < 5%, absence of circulating blasts, absence of extramedullary disease, absolute neutrophil count (ANC) >= 1,000/uL, platelet count > 100,000/uL
  * Complete remission with incomplete hematologic recovery (CRi), defined as all CR criteria except for residual neutropenia (ANC < 1,000/uL) or residual thrombocytopenia (platelet count < 100,000/uL)
  * Morphologic leukemia-free state with adequate marrow recovery, defined as bone marrow blasts < 5%, ANC >= 500/uL, and platelet count >= 20,000/uL
* Minimal residual disease positive >= 0.01% based on MPFC

  * For participants in first remission, MRD positivity at any point from time of establishing first remission onward while still in first remission
  * For participants in second remission, MRD positivity at any point from time of establishing second remission onward while still in second remission
  * MRD must be repeated and remain positive if additional treatment is given prior to enrollment
* CD123 positivity on flow cytometry (partial, dim, or bright) from either:

  * Conventional flow cytometry on marrow specimen from time of original diagnosis or first relapse
  * High-sensitivity multiparametric flow cytometry on marrow specimen from time of MRD positivity
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Serum albumin level >= 3.2 g/dL in the absence of receiving albumin infusion
* Serum total bilirubin =< 1.5 mg/dL, unless considered due to Gilbert's disease or medication effect
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase =< 2.5 times the upper limit of normal, unless considered due to medication effect (eg, azole therapy)
* Creatinine clearance >= 60 mL/min based on Cockcroft-Gault glomerular filtration rate (GFR) and serum creatinine (Cr) =< 1.8 mg/dL
* Ability to give full informed consent
* Females of reproductive potential (postmenopausal for less than 24 consecutive months) must have a negative pregnancy test within 1 week of initiating treatment and may not be breastfeeding

Exclusion Criteria:

* MRD negativity < 0.01% at screening
* Intensive AML therapy within the past 14 days, or non-intensive targeted therapy within the past 7 days
* Cord blood as donor source
* Second malignancy that would be expected to limit survival within less than 2 years
* Cardiovascular disease that would result in high risk for toxicity, including:

  * Uncontrolled or New York Heart Association (NYHA) class III or VI congestive heart failure
  * Recurrent or uncontrolled angina
  * Unstable angina, myocardial infarction, or stroke in past 6 months
  * Uncontrolled hypertension
  * Arrhythmia not controlled by medication
* Left ventricular ejection fraction < 50%
* History of coronary stent placement that requires mandatory continuation of dual antiplatelet therapy
* Uncontrolled intercurrent illness that includes but is not limited to: uncontrolled infection, disseminated intravascular coagulation, psychiatric illness/compliance issues that would limit compliance with study protocol
* Any medical condition that in the opinion of the investigator places the participant at unacceptable risk for toxicity to investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-03 (Estimated); Primary Completion 2025-08-03 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Up to 42 days
  Grade >= 3 toxicity using Common Terminology Criteria for Adverse Events version 5.0 or severe persistent hematologic toxicity defined as absolute neutrophil count (ANC) < 500/uL OR platelet count < 10,000/uL in participants that have morphologic leukemia-free state (bone marrow blasts < 5%) are conditions for a dose limiting toxicity.

SECONDARY OUTCOMES:
Measurable residual disease (MRD) | At the end of cycle 1 and cycle 2 (each cycle is 28 days).
  As measured by the University of Washington multiparametric flow cytometry (MPFC) assay with sensitivity of 0.01%
MRD | Within 30 days prior to initiation of transplant conditioning regimen and at day 100 after transplant
  As measured by the University of Washington MPFC assay with sensitivity of 0.01%.
Number of days between investigational regimen day 28 and initiation of transplant conditioning regimen | Between investigational regimen day 28 and initiation of transplant conditioning regimen, through study completion, an average of 1 year.
Rate of sinusoidal obstruction syndrome | up to 1 year following investigational therapy
Relapse | Up to 1 year
  As defined by International Working Group criteria: the relapse rate and median duration of remission following allogeneic hematopoietic cell transplantation (HCT) will be reported along with an exact 95% confidence interval.
MRD progression | Up to 1 year
  Defined by presence of leukemia blasts >0.01% at any time after achieving MRD negativity (<0.01%).
Overall survival | 1 year after transplant
  Kaplan-Meier methods will estimate the overall survival at 1 year following allogeneic (allo)HCT. This analysis will be performed using the FAS. The 1-year survival estimate will be reported along with a 95% confidence interval.

OTHER OUTCOMES:
CD123 expression via immunohistochemical stain on leukemia blasts in the bone marrow specimen | at time of diagnosis or relapse and following cycle 1 and cycle 2 (each cycle is 28 days).
  CD123 expression, on the original bone marrow specimen at time of diagnosis or time of relapse and the bone marrow specimen at time of MRD negativity, will be described as bright, dim, partial, or negative; and summarized by mean, median, standard deviation, and interquartile range.
T-cell (CD3) chimerism via short tandem repeat assay | 30, 90, 180, and 365 days after transplant
  Days to achieve full T-cell chimerism following alloHCT will be characterized by Kaplan-Meier methods along with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Caspian Oliai, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Habtemariam,Bruck, Los Angeles, California
  - University of California San Francisco, San Francisco, California